CLINICAL TRIAL: NCT06275698
Title: HONEY for the Treatment of POst-Tonsillectomy Pain - a Double-blind, Randomised, Placebo Controlled, Single Site Trial
Brief Title: HONEY for the Treatment of POst-Tonsillectomy Pain
Acronym: HONEY-POT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: Manuka Doctor UK Ltd (Unknown); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RD2023-14 HONEY-POT; 323188 (Other: IRAS); 56974 (Other Grant/Funding Number: CPMS)
Record Dates: First submitted 2023-08-24; First posted 2024-02-23 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Post Surgical Pain; Analgesia
Keywords: Post-tonsillectomy pain; Tonsil surgery; Manuka honey; Honey
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Alginates; Flavoring Agents

STUDY DESIGN:
Intervention Model Description: Intervention arm - Manuka honey, to be taken per-oral 15ml TDS for 14 days post-tonsillectomy.
  Placebo - sugar-based syrup, thickened with sodium alginate and with honey flavouring, to be taken per-oral 15ml TDS for 14 days post-tonsillectomy.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Intervention (Manuka honey) and placebo will be supplied in identical opaque jars with identical labels apart from individual unique ID numbers to facilitate un-blinding in the case of adverse events.
  Neither the patient nor the researcher collecting data will be aware of which arm the patient has been enrolled onto.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Manuka honey, 15ml, three times a day, for 14 days. To be kept on the tongue for at least 10 seconds prior to swallowing.
  Interventions: Dietary Supplement: Manuka honey MGO 1000
- Placebo (Placebo Comparator): Sugar-based syrup, thickened with sodium alginate and flavoured with honey flavouring, 15ml, three times a day, for 14 days.
  To be kept on the tongue for at least 10 seconds prior to swallowing.
  Interventions: Dietary Supplement: Sugar-based syrup, thickened with sodium alginate and flavoured with honey flavouring

INTERVENTIONS:
Dietary Supplement: Manuka honey MGO 1000 — Natural Manuka honey, produced in New Zealand. With MGO content ≥ 1000.
  Arms: Treatment
Dietary Supplement: Sugar-based syrup, thickened with sodium alginate and flavoured with honey flavouring — Sugar-based syrup, thickened with sodium alginate and flavoured with honey flavouring, 15ml, three times a day, for 14 days.
  To be kept on the tongue for at least 10 seconds prior to swallowing.
  Arms: Placebo

SUMMARY:
Double-blind, randomised, placebo controlled, single-site trial in adults to compare the effect of Manuka honey with standard of care compared to placebo with standard of care on post-tonsillectomy pain and postoperative outcomes.

Main aim is to investigate a potential improvement in post-tonsillectomy pain control, with a low cost and freely available alternative to conventional analgesics. Recent systematic review and multidisciplinary consensus suggest a potential role for the inclusion of honey for this purpose. Clinical efficacy over placebo remains to be conclusively demonstrated in robust clinical trials.

DETAILED DESCRIPTION:
Tonsillectomy is one of the most common surgical procedures performed in the UK. It can be a painful operation to recover from, particularly in adults. Amongst the recognised complications, poor oral intake secondary to uncontrolled pain can result in re-admission to hospital, development of localized infection and subsequent bleeding. Post-operative analgesia regimes can vary depending on the individual surgeon preference or departmental policies, however generally it involves regular simple analgesics including paracetamol, ibuprofen and topical analgesic throat sprays or rinses. Commonly, opioid based analgesics such as codeine, tramadol and oramorph are needed in the post-operative period. Whilst these are generally effective, they can be associated with significant side effects such as constipation, drowsiness and nausea and prolonged use is not recommended.

Beehive products such as honey and propolis have been mentioned as wound dressings in ancient writings across the world, thousands of years before the advent of modern medicine. Honey is a by-product of flower nectar produced in the aero-digestive tract of bees and propolis is produced from plant resins, enriched with salivary enzymatic secretions. Honey has been shown to possess anti-bacterial and anti-inflammatory properties. Manuka honey is a mono-floral honey with potential wound repair and antibacterial activities. It is produced by bees fed on the flowers of the New Zealand Manuka bush (Leptospermum scoparium) and contains a significantly higher concentration of the 1,2-dicarbonyl compound methylglyoxal, which may account for its antibacterial activity. Manuka honey has been reported to stimulate the formation of new blood capillaries and the growth of fibroblasts and epithelial cells when applied topically to wounds. It is now part of the routine armamentarium of products used in the treatment of burns and external skin wounds in NHS Plastic surgery departments in the United Kingdom (UK). The clinical efficacy of Manuka honey in the oral and oropharyngeal cavities is controversial and quality, placebo controlled, randomized clinical trials are lacking. There are a number of systematic reviews that have described some benefit of Manuka honey in the treatment of radiation induced oro-mucositis, particularly in reducing treatment interruptions, preventing weight loss and pain control.

The most recent PROSPECT (Procedure-specific postoperative pain management) guideline for tonsillectomy published in 2021 in the Anaesthesia journal, represented an international, multidisciplinary collaborative effort providing recommendations on the most effective pain management following tonsillectomy. The fourth of five summative recommendations, based on systematic review of the current literature, is that analgesic adjuncts such as postoperative honey is recommended. Honey could provide significant improvements in post-operative pain scores as well as provide opioid-sparing benefits. This is a powerful mandate for further research into the routine clinical usage of honey as an adjunct to post-tonsillectomy pain management. To date there have not been any placebo controlled, randomised clinical trials comparing the effectiveness of oral honey in post-tonsillectomy pain control in the UK.

The aim of this double-blind, randomised, placebo controlled clinical trial is to compare the effect of Manuka honey with standard of care compared to placebo with standard of care on post-tonsillectomy pain and postoperative outcomes. The hypothesis is that the addition of Manuka honey to standard of care will result in a significant reduction in post-tonsillectomy pain scores compared to the placebo control. The null hypothesis is that there is no significant difference between Manuka honey compared to placebo in post-tonsillectomy pain scores.

The primary endpoint/outcome are daily pain scores measured via Visual Analogue Scale (VAS). This is a continuous variable, which will be measured and recorded three times a day, every day for the first 14 days post-tonsillectomy.

The secondary endpoint/outcomes include the number and frequency of concurrent analgesia usage, the rate of readmission to hospital, the rate of secondary haemorrhage, the rate of infection requiring antibiotics treatment, the speed of return to work. These are a mixture of continuous and ordinal variables and will be collected retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18years old at the time of giving consent)
* Consented and listed for bilateral tonsillectomy or adenotonsillectomy
* Tonsillectomy performed within the trial study period

Exclusion Criteria:

* Any concurrent Head & Neck (H&N) malignancy
* Unilateral tonsillectomy
* Pregnancy
* Concurrent pharyngeal or upper aerodigestive tract biopsy
* Robotic tonsillectomy
* Previous H&N malignancy
* Previous H&N radiotherapy
* Type 1/2 diabetes mellitus
* Known allergy to bee related products
* Known allergy to golden syrup
* History of chronic pain
* History of fibromyalgia
* Current usage of chronic (>6weeks) analgesia
* High-risk anaesthetic patients
* Children or adolescents <18years old
* Adults unable to consent for themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-09-04 (Estimated); Study Completion 2025-09-04 (Estimated)

PRIMARY OUTCOMES:
VAS pain scores | 14 days post-tonsillectomy
  Pain scores as measured on a visual analogue scale 1-10.This is a continuous variable, which will be measured and recorded three times a day, every day for the first 14 days post-tonsillectomy.

SECONDARY OUTCOMES:
Number and frequency of concurrent analgesia usage | 14 days post-tonsillectomy
  Patients will be asked record their analgesia administration at home.
Rate of readmission to hospital | 14 days post-tonsillectomy
  Retrospective record of re-admission rate
Rate of secondary haemorrhage | 14 days post-tonsillectomy
  Retrospective record of secondary haemorrhage rate, defined as any haemorrhage after 24hrs post surgery
Rate of infection requiring antibiotics treatment | 14 days post-tonsillectomy
  Retrospective record of any related infection requiring antibiotic treatment
Speed of return to work | 14 days post-tonsillectomy
  Recording how quickly the patient is able to return to their normal occupation responsibilities

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Smith, PhD, Study Director — East and North Hertfordshire NHS Trust; George Mochloulis, MD, Principal Investigator — East and North Hertfordshire NHS Trust
Locations (1):
- Lister Hospital, Stevenage, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aldamluji N, Burgess A, Pogatzki-Zahn E, Raeder J, Beloeil H; PROSPECT Working Group collaborators*. PROSPECT guideline for tonsillectomy: systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2021 Jul;76(7):947-961. doi: 10.1111/anae.15299. Epub 2020 Nov 17. PMID 33201518
- [Background] Nolan VC, Harrison J, Wright JEE, Cox JAG. Clinical Significance of Manuka and Medical-Grade Honey for Antibiotic-Resistant Infections: A Systematic Review. Antibiotics (Basel). 2020 Oct 31;9(11):766. doi: 10.3390/antibiotics9110766. PMID 33142845
- [Background] Carter DA, Blair SE, Cokcetin NN, Bouzo D, Brooks P, Schothauer R, Harry EJ. Therapeutic Manuka Honey: No Longer So Alternative. Front Microbiol. 2016 Apr 20;7:569. doi: 10.3389/fmicb.2016.00569. eCollection 2016. PMID 27148246
- [Background] Hawley P, Hovan A, McGahan CE, Saunders D. A randomized placebo-controlled trial of manuka honey for radiation-induced oral mucositis. Support Care Cancer. 2014 Mar;22(3):751-61. doi: 10.1007/s00520-013-2031-0. Epub 2013 Nov 13. PMID 24221577
- [Background] Yang C, Gong G, Jin E, Han X, Zhuo Y, Yang S, Song B, Zhang Y, Piao C. Topical application of honey in the management of chemo/radiotherapy-induced oral mucositis: A systematic review and network meta-analysis. Int J Nurs Stud. 2019 Jan;89:80-87. doi: 10.1016/j.ijnurstu.2018.08.007. Epub 2018 Aug 23. PMID 30352321
- [Background] Cho HK, Jeong YM, Lee HS, Lee YJ, Hwang SH. Effects of honey on oral mucositis in patients with head and neck cancer: A meta-analysis. Laryngoscope. 2015 Sep;125(9):2085-92. doi: 10.1002/lary.25233. Epub 2015 Mar 16. PMID 25778825